CLINICAL TRIAL: NCT07329426
Title: Effects of Muscle Energy Technique Combined With Mobilization in Patients With Sacral Torsion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/24
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sacral Torsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maitland Mobilization With Muscle Energy Technique (PFS) (Experimental): Participants in this group will receive Maitland mobilization technique, two sets of 60 oscillations for 30 seconds, directed at sacrum according to standard graded oscillatory movements, grade 1 or 2 in week 1 and grade 3 or 4 in week 2. Muscle Energy Technique (MET) will also be applied to this group targeting specific muscles contributing to sacral torsion (e.g., piriformis, hamstrings, quadratus lumborum), with the purpose of correcting asymmetry, improving joint alignment, and enhancing the overall effectiveness of mobilization. The contract time will be 6-10 seconds and Hold time will be 15 seconds.
  Interventions: Procedure: Muscle Energy Technique + Maitland Mobilization
- Maitland Mobilization (Experimental): Participants in this group will receive Maitland mobilization technique, two sets of 60 oscillations for 30 seconds, directed at the sacrum. Mobilization will be applied according to the standard graded oscillatory movements grade 1 or 2 in week 1 and grade 3 or 4 in week 2, aiming to restore joint mobility, reduce pain, and improve function. No additional interventions will be provided.
  Interventions: Procedure: Maitland Mobilization

INTERVENTIONS:
Procedure: Muscle Energy Technique + Maitland Mobilization — Group A will receive Muscle energy technique with Maitland mobilization. Treatment protocol given to both groups will be carried out for 3 sessions per week for 2 weeks.
  Post Facilitation Muscle Energy Technique. WEEK 1:
  * Hot pack (10 minutes)
  * Post-Facilitation MET for piriformis, Quadratus Lumborum and Hamstrings.
  WEEK 2:
  * Hot pack (10 minutes)
  * Post-Facilitation MET for piriformis, Quadratus Lumborum and Hamstrings.
  Arms: Maitland Mobilization With Muscle Energy Technique (PFS)
Procedure: Maitland Mobilization — Group B will not receive any form of Muscle Energy Technique (MET). Instead, the intervention will consist exclusively of a joint mobilization technique directed at Sacrum.
  Arms: Maitland Mobilization

SUMMARY:
Project Summary Low Back Pain is one of the most prevalent musculoskeletal conditions worldwide. More than 70% of the people experience low back pain at some time in their life. The sacroiliac joint has been found to be the source of pain in 30% of mechanical low back pain sufferers. Sacral torsion is one of the types of SIJ dysfunction. This randomized controlled trial, conducted at Fauji Foundation Hospital and Foundation University College of Physical Therapy will assess the effects of combining muscle energy technique with mobilization on pain, lumbar range of motion, disability and active straight leg raise. Participants will be randomly assigned to either mobilization alone or mobilization with muscle energy technique, performed three times per week for two weeks. Data will be collected at baseline and at end of study (week 2) using the Numeric pain rating scale, goniometer, inclinometer and oswestry disability index. This study addresses a research gap by exploring combined effects of muscle energy technique (PFS) and Maitland mobilization for sacral torsion in improving pain, lumbar mobility, disability and active straight leg raise.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal conditions globally, with over 70% of individuals experiencing it at some point in their lifetime. It is the leading cause of disability worldwide and remains the primary global contributor to years lived with disability. A significant source of mechanical low back pain is the sacroiliac joint (SIJ), which accounts for 15% to 30% of cases, making it a key area of interest in both diagnosis and treatment.

SIJ dysfunction typically presents with localized pain and stiffness and can be difficult to differentiate from other causes of LBP such as lumbar spine or hip pathology. The dysfunction usually results from abnormal joint motion or malalignment, often linked to repetitive stress or minor subluxation that damages the joint capsule or posterior ligamentous structures. SIJ dysfunction can be categorized into five main types: anterior rotation, posterior rotation, up slip, down slip, and sacral torsions.

Sacral torsions are a specific type of SIJ dysfunction involving asymmetrical movement of the sacrum along a physiologic oblique axis, leading to joint fixation. These torsions are commonly described in osteopathic literature and include four types: Left-on-Left, Right-on-Right (forward torsions), and Right-on-Left, Left-on-Right (backward torsions). Such dysfunctions are frequently associated with asymmetries in lumbo-pelvic rhythm, leg length discrepancies, scoliosis, and muscular imbalances, particularly involving the hamstrings, piriformis, and quadratus lumborum. These biomechanical and muscular irregularities contribute to pelvic asymmetry during functional movements like forward flexion.

Muscle imbalances play a crucial role in the development and persistence of SIJ dysfunction. These may arise from adaptive responses or underlying biomechanical issues, leading to altered motor control and impaired movement quality. Balance in muscle strength and length, especially between corresponding groups on the left and right sides, is essential for maintaining proper pelvic alignment. Studies such as Jacobs et al. (2005) have shown significant asymmetries in hip abductor strength, highlighting the importance of bilateral symmetry in functional movement.

Conservative management of chronic SIJ dysfunction commonly includes physical therapy, manual therapy, activity modification, and pharmacological interventions such as analgesics and anti-inflammatory medications. Among manual therapy techniques, Muscle Energy Technique (MET) is widely used to address muscle imbalances by utilizing voluntary isometric contractions to engage autogenic or reciprocal inhibition mechanisms. This process activates the Golgi tendon organs, reducing muscle tension and facilitating improved joint mobility. A variation of MET, known as Post-Facilitation Stretch (PFS), involves a maximal isometric contraction followed by a rapid stretch, and has been shown to effectively increase flexibility and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 22- 44 years (18)
* Both males and females
* Clinically diagnosed sacral torsion. (Annexure E)
* Patients with pain intensity of at least 5 on NPRS
* Positive standing flexion test
* Positive seated flexion test
* Positive Gillet test
* Uneven anatomical landmarks (Sacral Sulcus, Inferior Lateral Angle, Lumbar Lordosis, Lumbar scoliosis, L5 position)

Exclusion Criteria:

* 1. Neurological deficits (hemiparesis, paralysis) 2. Pregnancy 3. Spinal surgery of any kind 4. Antero-Retro Spondylolisthesis diagnosed through radiological findings 5. Degenerative disc disease diagnosed through radiological findings 6. Spinal stenosis 7. Infection, tumors, osteoporosis, spinal fracture

Ages: 22 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  n=Numeric Pain Rating Scale (NPRS) will be used, 0 means no pain and 10 means worst pain.
Functional Disability | 2 weeks
  Oswestry Disability Index
Lumbar Mobility | 2 weeks
  Inclinometer will be used for checking the lumbar mobility
Active Straight Leg Raise | 2 weeks
  Goniometer will measure Active Straight Leg Raise

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan